CLINICAL TRIAL: NCT06276036
Title: Autoimmune Cytopenias as a Sign of Primary Immunodeficiency: Immunological and Molecular Approach to Optimize the Diagnostic-therapeutic Pathway
Brief Title: Autoimmune Cytopenias as a Sign of Primary Immunodeficiency.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Eleonora Gambineri, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAPID
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Cytopenia
MeSH Terms: conditions — Cytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Identification of specific markers (Experimental): Analysis of the immunological profile, Genetic analysis using next-generation sequencing (NGS) technology, Bioinformatic analysis, Functional studies.
  Interventions: Other: Identification of specific markers

INTERVENTIONS:
Other: Identification of specific markers — Analysis of the immunological profile, Genetic analysis using next-generation sequencing (NGS) technology, Bioinformatic analysis, Functional studies.

SUMMARY:
Autoimmune cytopenias resistant to treatment are among the most common clinical manifestations observed in patients with congenital alterations of the immune system, such as primary immunodeficiencies (PI). The exact contribution of immune system alterations to the pathogenesis of autoimmune cytopenias has not yet been fully elucidated. Moreover, conventionally employed therapeutic strategies often fail, leading to increased healthcare costs, high morbidity, and even mortality. Therefore, there is a need to establish clinical guidelines for diagnosis and to identify early biomarkers capable of identifying individuals responsive to therapy. Thus, a systematic approach to the study of such pathologies will allow for the identification of early biomarkers and facilitate the development of targeted therapeutic strategies

ELIGIBILITY:
Inclusion Criteria:

* Clinical and hematological diagnosis of autoimmune cytopenia

Additional inclusion criteria for classification into responder vs. non-responder:

* For immune thrombocytopenic purpura: platelet count increase >30,000 with at least a twofold increase from pre-treatment value
* For autoimmune hemolytic anemia: Hb ≥10 g/dL with an increase of at least 2 g/dL compared to baseline

Exclusion Criteria:

* Transient cytopenia without confirmation of autoimmunity where frontline treatment is not necessary

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of specific markers | Every three to six months
  The primary goal is to identify potential primary immunodeficiencies (PI) as responsible for autoimmune cytopenias through a comprehensive examination of clinical manifestations and the study of immune system cells in the patient cohort under investigation. The study will involve immunophenotypic investigation of T and B cell subsets using flow cytometry, the application of genomic approaches, and possibly the use of specific functional immunological tests to confirm and validate genetic results.

CONTACTS AND LOCATIONS:
Locations (6):
- University of South Florida, Tampa, Florida, United States
- Ghent University Hospital, Ghent, Belgium
- Italy (4):
  - Clinica Pediatrica - Università di Catania, Catania
  - Meyer Children's Hospital IRCCS, Florence
  - IRCCS Istituto Giannina Gaslini, Genova
  - Azienda Ospedaliero Universitaria Pisana, Pisa

IPD SHARING:
Plan to Share IPD: No